CLINICAL TRIAL: NCT06798857
Title: Exploration of the Relationship Between Mismatch Repair Status of Colorectal Cancer and Lymph Node Metastasis Patterns and Pathological High-risk Factors
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cai Zerong, Deputy Chief Physician, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2024ZSLYEC-289
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The pathological specimens before operation and the specimens after operation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pMMR group: Pathological immunohistochemical results suggested pMMR
- dMMR group: Pathological immunohistochemical results suggested dMMR

SUMMARY:
This study analyzed the differences in clinical baseline features and survival outcomes between pMMR and dMMR patients. The aim is to evaluate the impact of MMR status on overall survival and disease-free survival of colorectal patients, and to explore the population exempt from extended resection, so as to provide evidence-based medical evidence for the relationship between MMR status, lymph node metastasis pattern and clinicopathological risk factors in colon cancer patients.

DETAILED DESCRIPTION:
In recent years, colorectal cancer has become one of the most common cancers worldwide, and its prevalence and mortality are among the top three malignant tumors . Mismatch repair protein is considered to be one of the risk factors affecting the development of colorectal cancer, including MSH2, MSH6, MLH1, PMS2 and so on. However, their exact relationship to lymph node metastasis in patients with colorectal cancer is unclear. Studies have found that loss of expression of mismatch repair protein and positive expression of Her-2 are associated with lymph node metastasis in patients with colorectal cancer. On the other hand, MSI-H/dMMR colorectal cancer patients have a similar set of pathological features , such as the right half colon is more common, and lymph node or distant organ metastasis is less, but the relationship between the loss of mismatch repair status and skipping lymph node metastasis and other factors such as cancer nodules, nerve tract infiltration, and vascular cancer embolus has been ignored.

Right hemicolectomy combined with regional lymph node dissection is the standard operation for right hemicolectomy.However, there is no consensus on the scope of dissection, and different guidelines put forward different recommendations. For example, complete mesocolic excision (CME) combined with central vessel ligation (CVL) is recommended in Europe and the United States, while D3 surgery proposed by Japan has a large surgical risk. The surgical practice in China is consistent in principle with CME, but the scope of lymph node dissection tends to follow the Japanese D2/D3 scope of dissection, resulting in the lack of uniform standard.

Some studies have shown that expanding the scope of lymph node dissection can reduce the risk of local recurrence and distant metastasis, but this advantage is more significant in stage I to II patients, and there is no statistical difference in stage III colon cancer. At the same time, some studies have questioned the necessity of D3 dissection, arguing that the central group of lymph node metastasis is not significant, so D3 dissection is an overtreatment.

Therefore, the relationship between MMR status, lymph node metastasis pattern and clinicopathological risk factors in colon cancer patients needs to be further studied. Such research helps to stratify the management of patients at different risks and develop the most effective lymphatic dissection program for them, so as to provide individual and most appropriate treatment for each patient, in order to achieve the best treatment outcome and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* The preoperative diagnosis was primary colon adenocarcinoma;
* Undergoing radical surgical treatment;
* Postoperative immunohistochemistry to determine MMR status;
* Having complete key clinical and follow-up data.

Exclusion Criteria:

* Previous history of malignant tumors
* Concurrent distant metastasis
* Receiving preoperative neoadjuvant therapy.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects were colon cancer patients who received radical surgical treatment at the Sixth Affiliated Hospital of Sun Yat-Sen University from January 2010 to December 2021. Patients must not have received neoadjuvant chemoradiotherapy and have a clear MMR status and necessary clinical and pathological information as well as follow-up prognostic information
Sampling Method: Non-Probability Sample
Enrollment: 1471 (Actual)
Dates: Start 2009-04-14 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
DFS | From the date of the initial surgery to death or disease recurrence or metastasis,assessed up to 120 months
  Disease Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Zerong Cai, MD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Please contact us by Email